CLINICAL TRIAL: NCT04063540
Title: Acid-Sensing Ion Channel and Migraine Disease Proof of Concept Study on the Efficacy of Amiloride in the Prophylaxis of Migraine Aura
Acronym: APAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16-API-01
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Migraine With Aura
Keywords: migraine; aura; Amiloride; acid-sensing ion channel
MeSH Terms: conditions — Migraine with Aura; Migraine Disorders; Epilepsy | interventions — Amiloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo-amiloride (Other): Patients will be treated for 12 weeks with placebo and then after a 4 week wash-out period, will be treated for 12 weeks with amiloride.
  Interventions: Drug: Amiloride; Drug: Placebos
- amiloride -placebo (Other): Patients will be treated for 12 weeks with amiloride and then after a 4 week wash-out period, will be treated for 12 weeks with placebo.
  Interventions: Drug: Amiloride; Drug: Placebos

INTERVENTIONS:
Drug: Amiloride — Treatment by Amiloride vs placebo in crossover
Drug: Placebos — Treatment by Amiloride vs placebo in crossover

SUMMARY:
Recent data suggest involvement of Acid-Sensing Ion Channel channels in the pathophysiology of migraine making these channels a therapeutic target of migraine disease. The implication of Acid-Sensing Ion Channels is discussed through Acid-Sensing Ion Channel-1 which is the most expressed Acid-Sensing Ion Channel channel subtype in the central nervous system. In a mouse model, cortical spreading depression is inhibited by different Acid-Sensing Ion Channel blockers including amiloride which is a non-selective blocker of the Acid-Sensing Ion Channel-1 channel. From a translational perspective, an efficacy of amiloride on a series of migraine patients suffering from severe aura in open conditions. The APAM study is a proof-of-concept study that aims to evaluate the effect of amiloride in the prophylaxis of migraine with aura. This is a randomized crossover study versus placebo conducted in 3 French headache centers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine with aura code
* At least 1 aura with aura per month in the 3 months prior to inclusion
* No prophylactic antimigraine treatment for at least 1 month prior to inclusion
* For women of childbearing age, use of a reliable contraceptive method at least 3 months before and 1 month after the study
* Signature of written informed consent
* Patient affiliated with Social Security

Exclusion Criteria:

* Existence of contraindication to taking amiloride:

  * Known hypersensitivity to the molecule
  * Hyperkalemia (potassium level (> 5.5 mmol / l))
  * Use of another hyperkalemic diuretic or potassium salts
  * Renal insufficiency (clearance <60 ml / min)
  * Severe hepatocellular insufficiency
  * In combination with lithium, converting enzyme inhibitors, angiotensin II inhibitors (except if there is hypokalemia), ciclosporin, tacrolimus, non-antiarrhythmic drugs giving torsades de pointes
* Cardiovascular and renal history, for subjects over 75 years old
* Patient, who from an investigator's point of view would not be compliant to the procedure of the study
* Pregnant or lactating patient
* Patient under trusteeship, under guardianship, protected by law

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of attacks with aura, with or without headache. | 12 weeks

SECONDARY OUTCOMES:
Number of days with migraine headache, with or without aura | 12 weeks
Functional repercussion | 12 weeks
  Anxiety and depression score on the Hospital Anxiety and Depression scale scale

CONTACTS AND LOCATIONS:
Overall Officials: Michel LANTERI-MINET, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (5):
- France (5):
  - Hôpital Pierre Wertheimer, Bron
  - CHU Gabriel Montpied, Clermont-Ferrand
  - AP-HM, Marly
  - CHU de Montpellier, Montpellier
  - CHU de NICE, Nice

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charles AC, Baca SM. Cortical spreading depression and migraine. Nat Rev Neurol. 2013 Nov;9(11):637-44. doi: 10.1038/nrneurol.2013.192. Epub 2013 Sep 17. PMID 24042483
- [Result] Ayata C, Jin H, Kudo C, Dalkara T, Moskowitz MA. Suppression of cortical spreading depression in migraine prophylaxis. Ann Neurol. 2006 Apr;59(4):652-61. doi: 10.1002/ana.20778. PMID 16450381
- [Result] Ligthart L, Boomsma DI, Martin NG, Stubbe JH, Nyholt DR. Migraine with aura and migraine without aura are not distinct entities: further evidence from a large Dutch population study. Twin Res Hum Genet. 2006 Feb;9(1):54-63. doi: 10.1375/183242706776403019. PMID 16611468